CLINICAL TRIAL: NCT00711425
Title: An Open, Prospective Study to Evaluate Implant Stability, Marginal Bone Adaptation and the Survival Rate of Astra Tech Dental Implant System, Fixture Osseospeed™, in Patients With Tooth Loss in the Posterior Mandible in an Early Loading Protocol.
Brief Title: Study on OsseoSpeed™ Implants in Patients Missing 2-5 Teeth in the Posterior Lower Jaw, Restored With Permanent Teeth Attached 6-7 Weeks Later
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YA-OSS-0002
Record Dates: First submitted 2008-07-07; First posted 2008-07-08 (Estimated); Results first posted 2011-09-26 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Jaw, Edentulous, Partially
Keywords: Jaw, Edentulous, Partially (posterior mandible)
MeSH Terms: conditions — Jaw, Edentulous, Partially; Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Device: OsseoSpeed™

INTERVENTIONS:
Device: OsseoSpeed™ — OsseoSpeed™, all dimensions

SUMMARY:
The purpose of the study is to evaluate Astra Tech Dental Implant System, Fixture Osseospeed™, in patients with tooth loss in the posterior mandible in an early loading protocol. Primary objectives are implant stability, marginal bone adaptation and survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* 18 years of age and over
* Edentulous in the posterior mandible, Kennedy class I or class II. Last natural tooth, or previously restored implant in function is canine or first bicuspid.
* Deemed by the investigator as likely to present an initially stabile implant situation suitable for early loading

Exclusion Criteria:

* Untreated caries and/or periodontal disease of residual dentition
* History of edentulism in the area of implant placement of less than two months
* Current need for pre-surgical bone or soft tissue augmentation in the planned implant area.
* History of pre-surgical bone or soft tissue augmentation, within12 months, in the planned implant area.
* Any systemic or local disease or condition that would compromise post-operative healing and/or osseointegration
* Need for systemic corticosteroids or any other medication that would compromise post-operative healing and/or osseointegration
* Present alcohol or drug abuse
* Unable or unwilling to return for follow-up visits for a period of 5 years
* Current use of smoking tobacco
* Pregnancy or lactation at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-02; Primary Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin A McGlumphy, D.D.S., Principal Investigator — The Ohio State University, College of Dentistry
Locations (3):
- United States (2):
  - The Ohio State University, College of Dentistry, Columbus, Ohio
  - University of Washington, Dept. of Restorative Dentistry, Seattle, Washington
- Georg-August-Universität, Göttingen, Abt. Mund-, Keifer-, und Gesicthschirurgie, Göttingen, Germany

REFERENCES:
- [Result] Schliephake H, Rodiger M, Phillips K, McGlumphy EA, Chacon GE, Larsen P. Early loading of surface modified implants in the posterior mandible - 5 year results of an open prospective non-controlled study. J Clin Periodontol. 2012 Feb;39(2):188-95. doi: 10.1111/j.1600-051X.2011.01816.x. Epub 2011 Nov 23. PMID 22111584

RESULTS

PARTICIPANT FLOW:
Groups:
- OsseoSpeed: Fixture Osseospeed Implants with diameter of 3.5, 4.0, 4.5 and 5.0 mm and lengths of 8, 9, 11, 13, 15 and 17 mm.
Period: Overall Study
Arm/Group | OsseoSpeed
Started | 45 (Implant placement in 45 patients. Implant loading (baseline) in 44 patients.)
Completed | 41
Not Completed | 4
Not completed — Protocol Violation | 1
Not completed — Death | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Per protocol analysis presented, this includes implants loaded 0 to 56 days from implant placement (134 implants in 44 patients).
Arm/Group | OsseoSpeed
Number analyzed (Participants) | 44
Age Continuous [Mean (Standard Deviation); unit: years] | 57 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 29
  Germany | 15

OUTCOME MEASURES:

1. Primary Outcome: Implant Survival Rate
Description: An implant that has failed to osseointegrate, lost its osseointegration or fractured will be considered a failure effective from the date of removal. The survival rate for individual implants will be analyzed at each visit. Cumulative implant survival rate will be calculated using Kaplan-Meier life-table estimation and reported as percentage of survived implants.
Time Frame: At 5 year follow-up
Population: as for baseline characteristics
Measure: Number; unit: Percentage of implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed
Number analyzed (Participants) | 44
Number analyzed (Implants) | 134
Percentage of implants | 100

2. Primary Outcome: Implant Stability
Description: Implant stability will be evaluated using Resonance Frequency Analysis (RFA). The RFA value is automatically translated into an Implant Stability Quotient index (ISQ), which runs from 1 to 100.
Time Frame: At 1 year follow-up
Population: Per protocol analysis presented, this includes implants loaded 0 to 56 days from implant placement (134 implants in 44 patients).At 1-year follow-up, 43 patients were still in the study and thus evaluable for the analysis.
Measure: Mean (Standard Deviation); unit: ISQ
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed
Number analyzed (Participants) | 43
Number analyzed (Implants) | 130
ISQ | 77.4 (7.1)

3. Primary Outcome: Marginal Bone Adaptation
Description: Marginal bone adaptation will be expressed as the distance from the implant reference point to the most coronal bone-to-implant contact on the mesial and distal side of the implant. Bone adaptation in millimeters at follow-up visit will be compared to values obtained Baseline (loading). Positive value indicates bone gain and negative value bone loss.
Time Frame: At 5 year follow-up
Population: Per protocol analysis presented, this includes implants loaded 0 to 56 days from implant placement (134 implants in 44 patients). At 5-year follow-up, 41 patients were still in the study and thus evaluable for the analysis.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed
Number analyzed (Participants) | 41
Number analyzed (Implants) | 123
Millimeter | -0.05 (1.96)

ADVERSE EVENTS:
Arm/Group | OsseoSpeed
Serious Adverse Events (participants affected / at risk) | 17/45
Other Adverse Events (participants affected / at risk) | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OsseoSpeed (N=45)
KIDNEY ABCESS (Renal and urinary disorders) | 1 (1)
LOWER LUMBAR PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
AORTIC ANEURYSM (Vascular disorders) | 1 (1)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
HEART ATTACK (Cardiac disorders) | 2 (2)
INTESTINAL PAIN (Gastrointestinal disorders) | 1 (1)
PT HAD MRI, CT SCAN + COLON OSCOPY DUE TO PAIN ON R ABDOMEN (Investigations) | 1 (1)
BACTERIAL LUNG INFECTION LED TO COLLAPSED LUNG (Respiratory, thoracic and mediastinal disorders) | 1 (1)
FLUID MASS REMOVED FROM LUNG AFTER INFECTION CLEARED (Surgical and medical procedures) | 1 (1)
HYSTERECTOMY (Surgical and medical procedures) | 1 (1)
HEART SURGERY (4 BYPASSES) (Surgical and medical procedures) | 1 (1)
TOXAEMIA AT RIGHT FOOT (Infections and infestations) | 1 (1)
INJECTIONS BECAUSE OF PAIN IN THE LUMBAR SPINE (Surgical and medical procedures) | 1 (1)
OPERATION, SECOND STENT (Surgical and medical procedures) | 1 (1)
CLEANSING OF FRONTAL SINUS (Surgical and medical procedures) | 1 (1)
CYSTECTOMIA, ABLATION OF WISDOM TEETH (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less